CLINICAL TRIAL: NCT06904963
Title: Efficacy of Oral Hygiene Instructions Carried Out Using an Intra-oral Scanner: a Randomized Controlled Trial
Brief Title: Efficacy of Oral Hygiene Instructions Carried Out Using an Intra-oral Scanner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Jacopo Lanzetti, Dental Hygienist, RDH, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000620
Record Dates: First submitted 2025-03-14; First posted 2025-04-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Oral Hygiene Education
Keywords: oral hygiene; Dental scan; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hygiene instruction with dental scan (Experimental): Patients are provided with education and motivation for home oral hygiene through the use of an intraoral scanner (Mach 2 - Mech & Human) with the creation of a digital model and with the aim of improving operator-patient communication.
  Interventions: Device: Motivation for oral hygiene through oral scanner
- Traditional oral hygiene instruction (No Intervention): Patients are provided with education and motivation for oral hygiene at home in a traditional way, through the use of a simple mirror.

INTERVENTIONS:
Device: Motivation for oral hygiene through oral scanner — The oral scanner is used to create a digital model of the patient's mouth with which the operator will provide personalized oral hygiene instructions.
  Arms: Oral hygiene instruction with dental scan

SUMMARY:
In the relationship between the dental hygienist and the patient, communication plays a key role in ensuring the quality of care, the patient's well-being, and adherence to oral hygiene recommendations. The professional must therefore consider the challenges and limitations of effective communication.

The dental hygienist is a healthcare professional who plays a crucial role in the prevention and promotion of oral health. These specialists assist and educate patients on oral hygiene practices. In order to communicate effectively, especially in today's modern society, it is essential to use increasingly advanced communication tools. The hygienist's task is to explore new technologies and communication methods to motivate patients.

Through empathetic, respectful, and personalized communication, a lasting relationship is often established between the hygienist and the patient. This is because their interactions are generally more frequent than those between the patient and the dentist. While professional oral hygiene sessions are recommended at least once a year for everyone, "fragile" patients-those with periodontal disease or other conditions-may require more frequent visits.

In everyday practice, it has been observed that patients tend to feel more comfortable discussing their doubts, concerns, and issues with dental hygienists rather than with dentists.

To achieve effective communication, various communication methods may be necessary. It will be interesting to determine whether technology can become a useful tool in dental hygienists' practice and positively influence patients' oral hygiene with long-lasting effects.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 80 years
* with good systemic health

Exclusion Criteria:

* Patients with conditions related to increased gingival bleeding
* Patients on drug therapy related to increased gingival bleeding
* Patients with cognitive and/or manual and/or sensory deficits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Plaque Control Record (PCR) | at least 62 days
  Presence of bacterial plaque on the tooth surface
Level of adherence to home oral hygiene procedures and devices | at least 62 days
  Evaluation of how well the patient follows the recommended home oral hygiene indications. The operator will give an evaluation from 1 (no adherence: the patient has not adopted the indications provided during the previous session) to 5 (total adherence: the patient has successfully adopted all the indications provided in the previous session) of the adherence demonstrated by the patient to the use of the devices and techniques of home oral hygiene.

SECONDARY OUTCOMES:
Full Mouth Bleeding Score (FMBS) | at least 62 days
  Percentage of bleeding gums: A higher percentage shows a worse situation of gum inflammation.
Level of concordance of home hygiene procedures and devices | at least 62 days
  Evaluation of how much the patient feels involved in the recommended home oral hygiene indications. The operator will give an evaluation from 1 (no concordance: the patient feels minimally involved in the procedures aimed at improving his home oral hygiene) to 5 (total concordance: the patient feels involved in all the procedures aimed at improving his home oral hygiene) of the concordance reported by the patient on the home oral hygiene procedures provided.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jung K, Giese-Kraft K, Fischer M, Schulze K, Schlueter N, Ganss C. Visualization of dental plaque with a 3D-intraoral-scanner-A tool for whole mouth planimetry. PLoS One. 2022 Oct 26;17(10):e0276686. doi: 10.1371/journal.pone.0276686. eCollection 2022. PMID 36288348
- [Result] Doi K, Yoshiga C, Kobatake R, Kawagoe M, Wakamatsu K, Tsuga K. Use of an intraoral scanner to evaluate oral health. J Oral Sci. 2021 Jun 29;63(3):292-294. doi: 10.2334/josnusd.21-0048. Epub 2021 Jun 9. PMID 34108300
- [Result] Willershausen B, Schlosser E, Ernst CP. The intra-oral camera, dental health communication and oral hygiene. Int Dent J. 1999 Apr;49(2):95-100. doi: 10.1111/j.1875-595x.1999.tb00515.x. PMID 10858739